CLINICAL TRIAL: NCT00684346
Title: A Pilot Study of 18FDG-PET Imaging to Detect Changes in Airways Inflammation in Cystic Fibrosis Patients After Treatment for a Pulmonary Exacerbation
Brief Title: 18FDG-PET Imaging to Detect Changes in Airways Inflammation in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Felix Ratjen, Division Head, Respiratory Medicine, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000011762
Record Dates: First submitted 2008-05-08; First posted 2008-05-26 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Cystic Fibrosis
Keywords: 18FDG-PET imaging; airway inflammation; cystic fibrosis; pediatric; pulmonary exacerbation
MeSH Terms: conditions — Cystic Fibrosis | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: 18-FDG

INTERVENTIONS:
Other: 18-FDG — The administered intravenous dose of 18-FDG is 0.14mCi/kg up to a maximum of 10mCi before each PET imaging scan is performed.

SUMMARY:
The purpose of this study is to determine if 18Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) imaging can detect changes in airways inflammation in Cystic Fibrosis (CF) patients after treatment for a pulmonary exacerbation.

DETAILED DESCRIPTION:
Neutrophils play a key role in the pathogenesis of CF lung disease. We know that neutrophilic inflammation is related to a decline in pulmonary function. Therefore, early anti-inflammatory intervention is an opportunity to slow this irreversible pulmonary destruction. However, the development of sensitive, non-invasive diagnostic tools of airways inflammation is essential to the study and implementation of anti-inflammatory therapies. Our current armentarium of measures of airways inflammation is limited. BAL is invasive and not clinically acceptable as a tool for the serial measurement of inflammation. Sputum samples are highly variable and not reliable.

18FDG-PET is a promising tool because it is non invasive, has been shown to quantify the amount and location of neutrophilic inflammation and has the potential to be used to track inflammation over time. Therefore, the goal of this research study is to evaluate the ability of 18FDG -PET imaging to detect changes in airways inflammation in CF patients in response to conventional treatment for a pulmonary exacerbation

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF as defined by two or more clinical features of CF and a documented sweat chloride > 60mEq/L by quantitative pilocarpine iontophoresis test or a genotype showing two well characterized disease causing mutations
* Informed consent and verbal assent (as appropriate) provided by the subject's parent or legal guardian and the subject
* Ages 6-18 and able to perform reproducible spirometry
* Admission to the Hospital for Sick Children for a pulmonary exacerbation

Exclusion Criteria:

* Inability to perform reproducible spirometry
* Diagnosis of Cystic Fibrosis Related Diabetes (CFRD)
* Medical instability that would preclude the ability to perform PET imaging
* FEV1% predicted < 40%
* The use of supplementary oxygen
* Pregnancy or breastfeeding
* Severe claustrophobia

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in airways inflammation detected by 18FDG -PET from baseline | Measured at end of treatment (day 14)

SECONDARY OUTCOMES:
Correlation of pre and post 18FDG-PET data with lung function (FEV1, FEF 25-75 and FVC), sputum neutrophil count and sputum free elastase | Measured at end of treatment (day 14)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- See also: Link to published study results — http://pubs.rsna.org/doi/10.1148/radiol.12111873?url_ver=Z39.88-2003&rfr_id=ori%3Arid%3Acrossref.org&rfr_dat=cr_pub%3Dpubmed&